CLINICAL TRIAL: NCT06833944
Title: Unraveling the Potential of Physical Activity in the Treatment of Familial Hypercholesterolemia: Impact of Exercise on Cardiorespiratory Fitness, Atherosclerosis Progression, and Underlying Mechanisms
Brief Title: High Intensity Interval Training in the Treatment of Familial Hypercholesterolemia (UPPA-FH)
Acronym: UPPA-FH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, José Antonio Vargas Hitos, José A. Vargas-Hitos, MD, PhD, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID2022-142844OB-I00
Record Dates: First submitted 2025-01-27; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Familiar Hypercholesterolemia
Keywords: Inflamation markers; Cardiovascular risk; Physical fitness; Exercise; Cardiovascular disease; LDL cholesterol
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Parallel group randomized and controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High Intensity Interval Training (HIIT) intervention program (Experimental): The HIIT protocol will involve 3 training sessions per week for 16 weeks (a total of 74 sessions lasting 36 minutes). The high-intensity intervals will follow the Norwegian 4 x 4-minute HIIT model: 4 bouts of 4 minutes of high intensity corresponding to a rating of perceived exertion (RPE) 15 to 18 on the Borg 6 to 20 Scale and an 85-95%HRmax, interspersed with 3-minute active recovery intervals (RPE of 11 to 13 and 54-69%HRmax).
  Interventions: Other: HIIT intervention program
- Moderate Intensity Continous Training (MICT) intervention program (Experimental): The MICT protocol will involve 3 training sessions per week for 16 weeks (a total of 74 sessions lasting 44 minutes). The workout will be performed at RPE 11 to 13 (54-69%HRmax) to provide an isoenergetic workload (same energy expenditure) as the HIIT group
  Interventions: Other: MICT intervention program
- Control group (No Intervention): The control group will follow a usual care regime during the intervention and will not participate in supervised exercise. However, the participants randomized to this group will be invited to participate in a similar intervention once the study is completed (waiting list control group).

INTERVENTIONS:
Other: HIIT intervention program — The HIIT protocol will involve 3 training sessions per week for 18 weeks (a total of 74 sessions lasting 36 minutes). The program will be divided into two phases: phase 1 (adaptation to HIIT training: during the first 4 weeks, the intensity will be progressively increased to ensure the safety and progressive physical conditioning of the patients.
  The high-intensity intervals will follow the Norwegian 4 x 4-minute HIIT model: 4 bouts of 4 minutes of high intensity corresponding to a rating of perceived exertion (RPE) 15 to 18 on the Borg 6 to 20 Scale33 and an 85-95%HRmax, interspersed with 3-minute active recovery intervals (RPE of 11 to 13 and 54-69%HRmax). This protocol has been widely applied and is safe in general and in clinical populations. Additionally, this protocol includes the training parameters recently proposed in a recent meta-analysis to maximize the training effects of HIIT on cardiorespiratory fitness (primary outcome).
  Arms: High Intensity Interval Training (HIIT) intervention program
Other: MICT intervention program — The MICT protocol will involve 3 training sessions per week for 18 weeks (a total of 74 sessions lasting 44 minutes). The workout will be performed at RPE 11 to 13 (54-69%HRmax) to provide an isoenergetic workload (same energy expenditure) as the HIIT group.
  Each session will include 3 parts: warm-up (5 min), main MICT workout (34 min), and a cool-down (5 min). Warm-up will include mobility, core, and aerobic exercise involving major muscle groups. The main workout (MICT) will include exercises involving major muscle groups using the same materials and rationale as commented on in the HIIT group. The cool-down phase will include aerobic exercise at a lower intensity, stretching, and relaxation exercises (RPE<11). The highest and average HR and RPE for each session will be registered.
  Arms: Moderate Intensity Continous Training (MICT) intervention program

SUMMARY:
This study has one main objective:

a) To assess the impact of two different supervised exercise interventions on cardiorespiratory fitness and markers of subclinical atherosclerosis in patients with Familiar Hipercolesterolemia (FH), and to unravel the underlying mechanisms behind these effects.

The starting hypothesis of the UPPA-FH project anticipates that both exercise interventions will produce a large increase in cardiorespiratory fitness and will improve significant markers of atherosclerosis in patients with FH, with high-intensity interval training program (HIIT) being more efficient than the moderate-intensity continuous training (MICT) modality. The main effects will be mediated by a significant change in the metabolomic signature of the participants. In addition, higher physical activity will be associated with more favorable markers of atherosclerosis progression, as shown through blood and image technique

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an inherited disorder characterized by high levels of LDL cholesterol and an increased risk of atherosclerosis and premature cardiovascular disease. From a clinical perspective, FH patients require lifelong management and monitoring of their cholesterol levels and may require multiple medications to control their cholesterol levels, leading to increased healthcare utilization and costs. From an economic perspective, the lifetime costs of managing FH can be significant and can include the cost of medications, diagnostic tests, and hospitalizations for cardiovascular events. In Spain, FH represents a heavy burden for the health care system, with direct costs of 37,299,000 €, indirect costs (due to loss of labor productivity) of 50,049,000 €, and an average of 25 years of life lost adjusted for labor productivity. From a public health perspective, FH affects around 25 million people worldwide that are at an increased risk of premature mortality, making FH a significant public health concern.

Hypercholesterolemia is one of the main vascular risk factors (VRF) related to the development of cardiovascular diseases (CVD), mainly myocardial infarction (MI) and stroke, the main causes of global mortality in the past decades. It is important to note that patients with FH present an increased prevalence of CVD at a very early age (44 years on average) and, in comparison to the general population, patients with FH have a 13.2 times higher risk of developing atherosclerotic CVD; specifically, up to 50% of men and 30% of women with FH will suffer an MI before the age of 60. Atherosclerosis is a complex process that involves endothelial dysfunction, inflammation, or oxidative stress. The presence of atherosclerosis can be assessed with positron emission tomography (PET), which has shown a high ability to predict the development of atherosclerotic plaque and cardiovascular events even after the consideration of classic VRF, so it is used as a method of early diagnosis of subclinical atherosclerosis in patients with chronic proinflammatory diseases. Therefore, the use of PET along with various plasma markers of inflammation in patients with FH (including C-reactive protein, [CRP], interleukin 10 [IL10], oxidized LDL [oxLDL], and the intracellular adhesion molecule 1 [ICAM1]), could allow the detection of atherosclerotic disease in the very early stages. Consequently, understanding novel markers that allow early identification of subclinical atherosclerosis, as well as strategies for reducing the VRF associated with FH, are key targets in these patients.

The treatment of hypercholesterolemia is primarily based on pharmacological therapies such as statins, ezetimibe, and monoclonal antibodies, which can decrease LDL cholesterol levels by up to 60%. However, the rate of achieving LDL cholesterol targets set by clinical practice guidelines is low (30-40%) due to poor tolerance to high doses of statins and other reasons. Importantly, new risk factors such as chronic vascular inflammation and oxidative stress are now considered in the etiology of atherosclerotic CVD beyond LDL cholesterol levels. Consequently, new treatment approaches are needed to address the treatment of FH as an important public health concern.

For all the above, unraveling the role of potential protective factors and interventions that might significantly improve the cardiometabolic profile and reduce the risk of morbi-mortality in this population, as well as the mechanisms involved, is of wide clinical and public health interest.

The UPPA-FH project will unravel the role of physical activity and different exercise interventions on critical health markers in men and women with FH and will study the mechanisms by which these effects are produced. For instance, whether the effects of exercise are mediated by changes in the metabolomic signature related to blood lipids will be explored. This will enable i) international institutions to develop clinical guidelines including exercise as a first-line treatment for the management of FH and ii) to unravel (for the first time) the potential mechanisms behind the effects of exercise in this population.

Physical activity and physical fitness are strong markers of health that are positively and strongly associated with survival in the general population and in patients with CVD. However, the role of physical activity on markers of atherosclerosis progression, inflammation, endothelial function, and other CVD risk factors in patients with FH has not been explored and would provide a framework for targeted physical activity promotion interventions. Similarly, CRF is associated with a better lipid profile, lower rates of pro-atherosclerotic VRF (hypertension, diabetes), and less subclinical atherosclerosis in different populations and is associated with a lower risk of death from all causes and a lower risk of death from cardiovascular diseases (CVD). CRF has also been shown to be a better predictor of mortality than other traditional vascular risk factors (VRF), such as hypercholesterolemia, hypertension, smoking, or type 2 diabetes. In men with hypercholesterolemia, higher cardiorespiratory fitness (CRF) is associated with up to 45% lower risk of CVD mortality, independent of other clinical risk factors, which underscores the importance of CRF in the primary prevention of CVD in patients with hypercholesterolemia. Therefore, exploring the value of CRF as a marker of health in patients with familial hypercholesterolemia (FH) and how exercise interventions can improve CRF is of high scientific and clinical value.

Although exercise interventions can reduce inflammation, oxidative stress and improve endothelial function in different populations and is a cost-effective therapy with similar benefits to pharmacological treatment in reducing CV and all-cause mortality, its effects in patients with FH have not been addressed before. The UPPA-FH will unravel the role of high-intensity interval training (HIIT) versus moderate-intensity continuous training (MICT) on cardiorespiratory fitness and the course of atherosclerosis in men and women with FH. These interventions have proved to be effective in improving CRF and improve CVD risk factors, and HIIT has been shown to be a time-efficient intervention that increases adherence due to the limited amount of time needed and the clinically relevant benefits in patients with and without CVD. HIIT protocols also improve anthropometric, metabolic, and vascular function in people with type 1 diabetes, type 2 diabetes, coronary disease, obesity, or the general population. Furthermore, HIIT has been shown to be safe in patients with high CV risk, such as those with coronary disease and heart failure, when developed in supervised environments.

Unlocking how physical activity and fitness impact the development of atherosclerosis and the unique metabolomic signature of men and women with FH is a key goal of this proposal. But we're not stopping there. The UPPA-FH project goes one step further to uncover the specific effects of different exercise interventions and regimens on key health markers for FH, such as cardiorespiratory fitness and atherosclerosis, and to understand the underlying mechanisms for these benefits. This proposal has the potential to make breakthrough discoveries that will pave the way for future interventions and for developing clinical guidelines, including exercise recommendations for FH patients, which are currently lacking.

The novelty of this proposal relies on discovering the extent to which exercise can improve key health parameters in FM patients, which is currently unknown. The clinical guidelines for these patients lack specific information on physical activity and exercise, which limits the ability of the health care system to benefit this population. Based on evidence on many similar populations, it can be affirmed that exercise has a huge potential to improve critical markers in patients with FH. Another novelty of the UPPA-FH study is to unravel the mechanisms underlying the effects of exercise, including inflammatory markers, oxidative stress and the metabolomic signature. Finally, also a novelty of this study will be to address the safety of moderate and high intensity exercise in this special population of high CV risk by providing detailed information about the adverse effects of the interventions; the lack of adverse effects reporting in exercise trials is a very common issue that this study will clearly address. All in all, through a highly collaborative y multidisciplinary research approach team and design, this study will contribute to improve the current management of FH patients, and will allow to understand the reasons why exercise is beneficial in this genetic condition.

ELIGIBILITY:
Inclusion criteria:

* Individuals with a diagnosis of genetic FH.
* > 18 years old.
* Minimum follow-up of 1 year in the Vascular Risk Clinic of the Virgen de las Nieves University Hospital (HUVN).
* Clinical and treatment stability.
* Non-pathological angio-TAC of coronary arteries in the 5 years prior to the study (for participants >45 years old).

Exclusion criteria:

* Inability to read, understand and sign the informed consent.
* Contraindications to exercise.
* History of clinical CVD (ischemic heart disease, stroke, and/or peripheral arterial disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Before and after the training intervention or control (16 weeks).
  It will be evaluated using the Bruce Protocol Ramp, variation of the most widely used protocol in cardiology units worldwide (Bruce Protocol). The test is performed on a treadmill, where the speed and incline will gradually increase every 15 seconds until exhaustion. Because CRF is the primary study outcome, the maximum oxygen uptake will be continuously measured with the Vyntus CPT (see budget). A 12-lead ECG will be used to monitor heart rhythm and blood pressure will also be monitored. The rating of perceived exertion (RPE, Borg scale 1-10), maximum heart rate (bpm at exhaustion) and recovery heart rate and blood pressure (1 and 3 minutes later, bpm) will be recorded.

SECONDARY OUTCOMES:
Vascular inflammation | Before and after the training intervention or control (16 weeks).
  Will be evaluated by performing a PET-CT. This examination is performed with an integrated PET/CT scanner (Siemens Biograph Vision 600, from Siemens Healthcare®, Erlangen, Germany). The protocol for the preparation procedure, administration of the radiopharmaceutical and image acquisition will be based on the available international recommendations. Before the examination, the patient is subjected to a fast of at least 6 hours and adequate hydration, and should present a capillary glucose level lower than 6.8 mmol/L (122.51 mg/dL) at the time of radiopharmaceutical administration. The evaluation of the images will include a visual and semi-quantitative analysis by calculating the different metabolic quantitative parameters that include the SUV (Standard Uptake Value) normalized by body weight and lean mass (SUL) maximum. The regions of interest (ROIs) for the calculation of SUL will be: carotid arteries, aortic arch, abdominal aorta and common iliac arteries.
Arterial Stiffness | Before and after the training intervention or control (16 weeks).
  Evaluated by determining the VOP, which depends on arterial stiffness (the more speed the more stiffness). Its elevation is a early marker of atherosclerosis. The Mobil-O-Graph® 24h pulse wave monitor device (IEM GmbH, Stolberg, Germany), whose operation is based on oscillometry recorded by a blood pressure cuff placed on the brachial artery, will be used.
Carotid Doppler Ultrasound | Before and after the training intervention or control (16 weeks).
  Non-invasive technique that allows visualization of the walls of the carotid artery using ultrasound. The General Electric's Logic F6® ultrasound device will be used, considering pathological both the presence of carotid plaque and an intima-media thickness (IMT) greater than >0.9 mm, both markers of subclinical atherosclerosis.
Physical activity | Before and after the training intervention or control (16 weeks).
  This important variable for the study will be assessed with triaxial accelerometers (Axivity AX3, Axivity Ltd, United Kingdom) to characterize the physical activity status during approximately 10 days. The AX3 has been validated and used to measure physical activity in a previous large-scale cohort study. Participants will use the accelerometer on the non-dominant wrist 24 hours a day for 10 consecutive days. A sampling frequency of 25 Hz will be set. Unprocessed accelerometry data will be downloaded as ".cwa" files and processed with R software using the GGIR package (v. 2.5-0, https://cran.r-project.org/web/packages/GGIR/)39. The most current thresholds will be applied to calculate the amount of time in sedentary activities, light, moderate, vigorous and very vigorous activities.
Diet | Before and after the training intervention or control (16 weeks).
  Adherence to mediterranean diet will be evaluated using the PREDIMED questionnaire.
Ultrasensitive PCR | Before and after the training intervention or control (16 weeks).
  Inflammatory marker (mg/L).
IL-6 | Before and after the training intervention or control (16 weeks).
  • Inflammatory marker: (pg/mL).
IL-10 | Before and after the training intervention or control (16 weeks).
  Inflammatory marker: (pg/mL).
Oxidized LDL | Before and after the training intervention or control (16 weeks).
  Oxidative stress marker: (U/L)
ICAM-1 | Before and after the training intervention or control (16 weeks).
  Endothelial dysfunction marker: (pg/mL)
Vitamin D | Before and after the training intervention or control (16 weeks).
  Parameter involved in muscle metabolism: (nmol/L).
TSH | Before and after the training intervention or control (16 weeks).
  Parameter involved in muscle metabolism (mUI/L).
Glucose | Before and after the training intervention or control (16 weeks).
  Glucose profile (mg/dL).
Triglycerides | Before and after the training intervention or control (16 weeks).
  Lipid profile (mg/dL).
Cholesterol | Before and after the training intervention or control (16 weeks).
  Total cholesterol (mg/dL), LDLc (mg/dL) and HDLc (mg/dL).
Apoproteins and lipoprotein a | Before and after the training intervention or control (16 weeks).
  Apoproteins and lipoprotein a.
Fibrinogen | Before and after the training intervention or control (16 weeks).
  Coagulation (mg/dL, von Clauss assay).
Homocysteine | Before and after the training intervention or control (16 weeks).
  Coagulation (μmol/l; AxSYM • Homocysteine; Abbott Laboratories, Abbott Park, IL).
Urea | Before and after the training intervention or control (16 weeks).
  Renal function (mg/dL).
Creatinine | Before and after the training intervention or control (16 weeks).
  Renal function (mg/dL).
Erythrocytes | Before and after the training intervention or control (16 weeks).
  Hemogram (x 106/uL).
Hemoglobin | Before and after the training intervention or control (16 weeks).
  Hemogram (Hb, g/dL).
Mean corpuscular volume | Before and after the training intervention or control (16 weeks).
  Hemogram (VCM, fL).
Leukocytes | Before and after the training intervention or control (16 weeks).
  Hemogram (x 103/uL).
Platelets | Before and after the training intervention or control (16 weeks).
  Hemogram (x 103/uL).
Microalbuminuria | Before and after the training intervention or control (16 weeks).
  Determination of albumin in urine by nephelometry (Hy-Pro 50 protein analyzer) (mg/dL).
Metabolites: Carbohydrates (glucose). | Before and after the training intervention or control (16 weeks).
  Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Metabolites: Amino Acids | Before and after the training intervention or control (16 weeks).
  Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Metabolites: Derivatives | Before and after the training intervention or control (16 weeks).
  E.g., 3-hydroxybutyrate, creatine. Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Metabolites: TCA cycle metabolites | Before and after the training intervention or control (16 weeks).
  E.g., citric acid, pyruvic acid. Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Metabolites: Choline | Before and after the training intervention or control (16 weeks).
  (Cho)-based compounds (which are essential components of cellular membranes). Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Metabolites: Nucleotides/nucleosides, polyols | Before and after the training intervention or control (16 weeks).
  E.g., glycerol. Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Metabolites: fatty acids and ketone bodies | Before and after the training intervention or control (16 weeks).
  E.g. 3-hydroxybutyrate, acetate, and acetoacetate. Acquisition of metabolomic profiles by Nuclear Magnetic Resonance (NMR) on a Bruker Avance Ascend HD 600 MHz spectrometer. The NMR profiles and other data will be analyzed by multivariate data analysis techniques to find relevant biomarkers and for the construction of predictive models. These analyses will be conducted at the University of Almería and a comprehensive lipidomic fingerprint will be performed by the BGI.inc in Hong Kong.
Upper body strength | Before and after the training intervention or control (16 weeks).
  Upper body strength will be evaluated using Hand Grip Strength (JAMAR dynamometer).
Lower body strength | Before and after the training intervention or control (16 weeks).
  Lower body strength will be evaluated using 30 Second Chair Stand Test.
Height | Before and after the training intervention or control (16 weeks).
  Height will be measured in cm with 1mm precision (SECA 222).
Weight | Before and after the training intervention or control (16 weeks).
  Weight will be measured in kg (SECA 222).
BMI | Before and after the training intervention or control (16 weeks).
  Weight will be measured in kg and height in cm with 1mm precision (SECA 222), and BMI will be calculated (in kg/m2).
Fat percentage | Before and after the training intervention or control (16 weeks).
  Total and localized fat percentage will be measured by densitometry (DEXA).
Muscle mass | Before and after the training intervention or control (16 weeks).
  Lean body mass and muscle mass will be measured by densitometry (DEXA).
Waist circunference | Before and after the training intervention or control (16 weeks).
  Waist circumference will be measured by non-elastic anthropometric tape (SECA 200).
Hip circumference | Before and after the training intervention or control (16 weeks).
  Hip circumference will be measured by non-elastic anthropometric tape (SECA 200).
Age | Before and after the training intervention or control (16 weeks).
  Years old.
Education Level | Before and after the training intervention or control (16 weeks).
  Categorical.
Occupational status | Before and after the training intervention or control (16 weeks).
  Categorical.
Family and personal history of CVD | Before and after the training intervention or control (16 weeks).
  Categorical.
Risk of suffering a cardiovascular event in 5 and 10 years | Before and after the training intervention or control (16 weeks).
  Will be estimated using the SAFEHEART-Risk Equation.
Anxiety | Before and after the training intervention or control (16 weeks).
  Self-perceived levels on anxiety will be evaluated using the HADS questionnaire.
Depression | Before and after the training intervention or control (16 weeks).
  Self-perceived levels on depression will be evaluated using the HADS questionnaire.
Individual Health | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life will be evaluated using the SF-36 questionnaire.
Physical Function | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life will be evaluated using the SF-36 questionnaire.
Physical Role | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (physical role) will be evaluated using the SF-36 questionnaire.
Pain | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (pain) will be evaluated using the SF-36 questionnaire.
General Health | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (general health) will be evaluated using the SF-36 questionnaire.
Vitality | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (vitality) will be evaluated using the SF-36 questionnaire.
Social Function | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (social function) will be evaluated using the SF-36 questionnaire.
Emotional Role | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (emotional role) will be evaluated using the SF-36 questionnaire.
Mental Health | Before and after the training intervention or control (16 weeks).
  Self-perceived levels of quality of life (mental health) will be evaluated using the SF-36 questionnaire.
Cognitive function | Before and after the training intervention or control (16 weeks).
  Cognitive function will be evaluated with the Montreal Cognitive Assessment (MoCA).
Working memory | Before and after the training intervention or control (16 weeks).
  Working memory will be evaluated with the National Institute of Health (NIH) Toolbox, a multi-domain neuropsychological test battery tests that are administered digitally. In particular, the List Sort Working Memory Test has been selected to define performance in working memory.
Visual and episodic memory | Before and after the training intervention or control (16 weeks).
  Visual and episodic memory will be evaluated with the National Institute of Health (NIH) Toolbox, a multi-domain neuropsychological test battery tests that are administered digitally. In particular, the Picture Sequence Memory Test has been selected to define performance in visual and episodic memory.
Cognitive flexibility | Before and after the training intervention or control (16 weeks).
  Cognitive flexibility will be evaluated with the National Institute of Health (NIH) Toolbox, a multi-domain neuropsychological test battery tests that are administered digitally. In particular, the Dimensional Change Card Sort Test has been selected to define performance in cognitive flexibility.
Inhibitory control and attention | Before and after the training intervention or control (16 weeks).
  Inhibitory control and attention will be evaluated with the National Institute of Health (NIH) Toolbox, a multi-domain neuropsychological test battery tests that are administered digitally. In particular, the Flanker Test has been selected to define performance in inhibitory control and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Vargas-Hitos, MD, PHD, Principal Investigator — Virgen de las Nieves University Hospital, Granada, Spain; Alberto Soriano Maldonado, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Virgen de las Nieves University Hospital, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided